CLINICAL TRIAL: NCT04386070
Title: Preventing Pulmonary Complications in Surgical Patients at Risk of COVID-19
Acronym: PROTECT-Surg
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of IMP availability - may resume.
Sponsor: University of Birmingham (Other)
Collaborators: Christian Medical College and Hospital, Ludhiana, India (Other); Ministry of Health, Ghana (Other Government); University of Lagos, Nigeria (Other); Kigali University Teaching Hospital (Other); Hospital Español Veracruz (Unknown); Université d'Abomey-Calavi (Other); University of Witwatersrand, South Africa (Other); University of Edinburgh (Other); Istituto Clinico Humanitas (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG_20-029 COVID-19; 2020-001448-24 (EudraCT Number)
Record Dates: First submitted 2020-04-30; First posted 2020-05-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Complications in Surgical Patients; COVID; Severe Acute Respiratory Syndrome
Keywords: Surgery; Pneumonia; COVID 19; COVID; SARS-Cov-2; SARS
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Pneumonia; COVID-19

STUDY DESIGN:
Intervention Model Description: The trial uses a Bayesian adaptive platform design, allowing for termination of arms if their superiority to standard care is established, and addition of new treatment arms. Patients will be randomised 1:1 to (A) Control (normal practice), (B) RESP301
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (normal practice) (No Intervention): Treatment without the trial intervention. Patients will be treated as per hospital routine practice. The control arm may change over the course of the trial and will be monitored by the TMG and DMC
- RESP301 (Experimental): RESP301 is administered quickly (8-10 minutes) via an easy-to-use, vibrating mesh nebuliser. The recommended nebulisers used to administer this intervention are available in all participating countries. The intervention will be administered using a nebuliser according to standard local practice; where permitted for patients to self-administer, a member of the clinical team will ensure that the patient has viewed the intervention administration training video, and will also oversee the patient for the first trial dose to ensure proper administration.
  Interventions: Drug: RESP301

INTERVENTIONS:
Drug: RESP301 — RESP301 is a formulation consisting of three agents already used in clinical practice: mannitol, sodium nitrite and citric acid. Delivered by a vibrating mesh nebuliser three times per day (TID) (at least 4 hours apart), for 7 days. Each dose of RESP301 is a 6ml admixture of 150mM NaNO2, 50mM mannitol and 100mM citric acid, buffered at pH 5.4.
  Arms: RESP301

SUMMARY:
The aim of this study is to reduce pulmonary complications in adult patients undergoing abdominal or thoracic surgery in COVID-19 exposed hospital environments. A Trial in Low and Middle Income Countries (LMICs)

DETAILED DESCRIPTION:
This trial has an adaptive platform design to identify at the earliest opportunity intervention arms which are showing benefit, drop arms which have a clear lack of benefit, and rapidly introduce new therapeutic options to the platform. This will enable rapid feedback of results to clinicians, allowing the standard of care to be modified as the pandemic progresses. Regular and frequent monitoring of results will be guided by an experienced, independent DMC.

Eligible patients will be randomised at the level of the individual in a 1:1 ratio between:

A. Control (normal practice) B. RESP301 6ml mixture of 150mM sodium nitrate, 50mM mannitol and 100mM citric acid, buffered at pH 5.4, three times per day (at least 4 hours apart), for 7 days or until discharge, whichever occurs first

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over. (This criteria MUST be made country-specific)
* Planned to undergo abdominal or thoracic elective or emergency inpatient surgery requiring general anaesthesia.
* Asymptomatic of COVID-19, including patients with: those not tested, negative test results, positive test but no symptoms (to be monitored post-surgery for symptoms)
* Informed patient consent.
* Able to operate a vibrating mesh nebuliser, as assessed by the recruiting physician

Exclusion Criteria:

* Procedures under local anaesthesia
* Known history of adverse reaction/contraindication to trial drug
* Pregnancy and/or lactating patients (including patients undergoing caesarean section)
* History of methaemoglobinaemia
* Patients receiving any type of prescribed nitric oxide-donating agents (e.g. Nitroprusside, Isosorbide dinitrate, Isosorbide mononitrate, Naproxcinod, Molsidomine and Linsidomine)
* Unable to tolerate use of a nebuliser and/or deemed unlikely to be able to adhere to protocol in view of investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6400 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Pneumonia free survival; acute respiratory distress syndrome (ARDS) free survival; or death | From randomisation until discharge from hospital, average less than 30 days
  The primary outcome is any one of the following, inpatient, postoperative pulmonary complications:
  Pneumonia Acute respiratory distress syndrome (ARDS) Death

SECONDARY OUTCOMES:
Rate of Pneumonia | From randomisation until discharge from hospital, average less than 30 days
  Pneumonia will be presented and analysed separately as a secondary outcome measure as well as within the composite primary outcome measure.
Rate of ARDs | From randomisation until discharge from hospital, average less than 30 days
  ARDs will be presented and analysed separately as a secondary outcome measure
Death rate | From randomisation until discharge from hospital, average less than 30 days
  Death will be presented and analysed separately as a secondary outcome measure
Rate of unexpected ventilation | From operation until 30 days post operation
  Unexpected inability to extubate and wean patient from ventilation after general anaesthesia, or reintubation and ventilation by 30 days after surgery
COVID-19 pulmonary complications | 30 days post-surgery
  Postoperative diagnosis of proven COVID-19 pulmonary complications
Duration of hospital stay | 30 days post-surgery
  Duration of hospital stay (including time spent in intensive care, time ventilated)
Pulmonary function | 30 days post-surgery
  Pulmonary function in keeping with the World Health Organisation (WHO) Solidarity Trial outcome scale

CONTACTS AND LOCATIONS:
Overall Officials: Aneel Bhangu, Principal Investigator — University of Birmingham
Locations (9):
- Nigeria (3):
  - University Of Abuja Teaching Hospital (Spoke), Gwagwalada
  - Lagos University Teaching Hospital (Hub), Lagos
  - Nnamdi Azikiwe University Teaching Hospital (Spoke), Nnewi
- Rwanda (6):
  - University Teaching Hospital of Butare (CHUB) (Spoke), Butare
  - Kibungo Referral Hospital (Spoke), Kibungo
  - Kibagabaga Hospital (Spoke), Kigali
  - University Teaching Hospital of Kigali (Hub), Kigali
  - Kibogora District Hospital (Spoke), Kirambo
  - Ruhengeri Referral Hospital (Spoke), Ruhengeri

IPD SHARING:
Plan to Share IPD: No
Hospital-level data will not be released or published. Country-level analyses will only be conducted with permission of lead investigators from each participating country. Local investigators may access their data across their country to perform country-level analyses (all participating hospitals should consent to their data being used in this way).

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343